CLINICAL TRIAL: NCT06938477
Title: EFFECTS OF THERA-TRAINER BASED EXERCISES ON MOTOR AND COGNITIVE PERFORMANCE AMONG HEMİPARATİC STROKE PATIENTS. A RANDOMİSED CONTROL TRİAL
Brief Title: Thera-Trainer Exercise Effects on Motor and Cognitive Outcomes in Stroke: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Fatma Kübra ÇEKOK, Asst.Prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: stroke; aerobic exercise; motor performance; cognitive performance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled study
Who Masked: Participant
Masking Description: Study participants are unaware of their assigned grou
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- THERA-TRAINER BASED EXERCISES (Experimental): Participants in the exercise arm will engage in structured, Thera-Trainer-based exercise programs tailored to their motor and cognitive rehabilitation needs. The intervention focuses on combining motor and cognitive tasks to maximize recovery outcomes.
  Interventions: Other: THERA-TRAINER BASED EXERCISES
- Functional Stroke Training (Experimental): To enhance motor recovery, functional independence, and cognitive performance in stroke patients
  Interventions: Other: FUNCTIONAL STROKE TRAİNİNG

INTERVENTIONS:
Other: THERA-TRAINER BASED EXERCISES — The interventions will carried out two days a week and 40 minutes for eight weeks
  Arms: THERA-TRAINER BASED EXERCISES
Other: FUNCTIONAL STROKE TRAİNİNG — he interventions will carried out two days a week and 40 minutes for eight weeks
  Arms: Functional Stroke Training

SUMMARY:
Technology-supported training supports the rehabilitation process by providing high-intensity, repetitive, and task-specific treatment, contributes to the recovery process, and facilitates the restoration of arm function (Bertani et al., 2017). Technology-supported rehabilitation studies for the upper extremity are performed using different devices. THERA-Trainer Tigo is used for the mobilization of individuals with limited mobility after trauma or due to any reason; it is suitable for passive movement training and active movement. Treatment with active-passive exercise devices facilitates rehabilitation with natural and rhythmic movements. It allows almost all patients, from wheelchair users to walkers, to actively participate in bicycle training during the rehabilitation process (Pazo et al., 2017). There are very few studies in the literature examining the relationship between cognitive and motor performance functions of THERA-Trainer-based exercises, and the aim of this study is to provide a preliminary idea in terms of progression to clinicians during the evaluation phase and treatment, to contribute to treatment, and to academic researchers.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability worldwide. It can be generally classified as ischemic stroke and hemorrhagic stroke. Ischemic stroke is defined as an infarction of the brain, spinal cord, or retina and accounts for approximately 70% of all strokes. Hemorrhagic stroke occurs as a result of intracerebral hemorrhage and subarachnoid hemorrhage (Campbell et al., 2019).Technology-assisted rehabilitation supports recovery by providing high-intensity, repetitive, and task-specific treatment, facilitating the restoration of upper limb function. Studies on technology-based rehabilitation for upper extremity recovery utilize various devices. The THERA-Trainer Tigo, for instance, is designed to mobilize individuals with restricted movement abilities caused by trauma or other conditions. It is suitable for both passive and active motion training. Therapy with active-passive exercise devices promotes rehabilitation through natural and rhythmic movements. It accommodates a wide range of patients-from wheelchair users to those capable of walking-by enabling nearly all individuals in the rehabilitation process to actively participate in cycling exercises .

However, there is a limited body of research exploring the relationship between cognitive and motor performance functions during THERA-Trainer-based exercises. This study aims to address this gap by providing clinicians with insights into progression during evaluation and treatment phases, enhancing therapeutic strategies, and contributing to the academic knowledge base for researchers.

ELIGIBILITY:
Inclusion Criteria:

* Having had an ischemic or hemorrhagic stroke for the first time
* Those with a Montreal Cognitive Assessment (MOCA) score above 21,
* Individuals with a functional level below 4 according to the modified Rankin scale (MRS),
* Individuals with upper extremity spasm below 3 according to the modified Ashword scale (MAS)

Exclusion Criteria:

* Montreal Cognitive Assessment (MOCA) score of less than 21,
* Upper extremity spasticy of over 3 according to MAS,
* Patients with subluxation and fracture risk in the shoulder,
* Agnosia or visual impairment,
* Limited joint movement in the hemiplegic side upper extremity,
* Patients who have undergone any botulinum toxin application or surgery in the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Mini Mental Test | Eight weeks
  The Mini Mental State Examination (MMSE) is a widely used tool for assessing cognitive function, particularly in screening for dementia and monitoring cognitive changes over time. It evaluates different cognitive domains, including orientation, registration, attention, calculation, recall, language, and visual-spatial skills.
Digit Span Test | Eight weeks
  The Digit Span Test is a cognitive assessment tool used to evaluate working memory, attention, and concentration. It is often part of broader neuropsychological evaluations and can assess both forward and backward digit span.
Frenchay Arm Test | Eight weeks
  The Frenchay Arm Test involves 5 tasks, each graded as pass (1 point) or fail (0 points) based on the patient's ability to complete the task. The tasks progress in difficulty and assess various aspects of upper limb function.
Time Up Go Test (TUG) | Eight weeks
  The Timed Up and Go Test (TUG) is a simple and widely used assessment tool to evaluate mobility, balance, and functional independence. It is particularly useful for identifying fall risk in older adults and individuals with neurological or musculoskeletal impairments.
Fugl Meyer Assesment | Eight weeks
  The test examines reflex activity, voluntary movements within, partially out and independent of synergies (22). The scale includes 33 items divided into 4 subscales: shoulder/elbow (A, 18 items), wrist (B, 5 items), hand (C, 7 items) and coordination/ speed (D, 3 items). Each item is scored on an ordinal 3-point scale, where 2 points are assigned when the movement is performed fully, 1 point when performed partially, and 0 points when the movement cannot be performed. A total score of 66 indicates better sensorimotor function
Five Time Sit to Stand | Eight weeks
  The Five Times Sit-to-Stand Test (FTSST) is a simple, reliable, and functional test used to assess lower limb strength, balance, and mobility. It is widely applied in clinical and research settings for evaluating physical performance in various populations, including older adults and individuals with neuromuscular conditions.The individual sits in a standard chair (seat height ~43-45 cm) without armrests.The chair is placed against a wall or a stable surface to prevent movement.The participant starts seated with their back against the chair and feet flat on the floor, arms crossed over the chest.On the signal "Go," they are instructed to stand up fully and sit back down as quickly as possible, repeating this motion five times.The test begins at the word "Go" and ends when the participant fully stands after the fifth repetition.A stopwatch is used to record the total time taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma KÜBRA Çekok, Tarsus, Mersin, Turkey (Türkiye)